CLINICAL TRIAL: NCT06130111
Title: Spatial Location of Breast Cancer Local Recurrence After Mastectomy: the Secret Study, a Retrospective Analysis.
Brief Title: Spatial Location of Breast Cancer Local Recurrence After Mastectomy
Acronym: Secret
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Albert Schweitzer Hospital (Other); Canisius-Wilhelmina Hospital (Other); Diakonessenhuis, Utrecht (Other); Erasmus Medical Center (Other); Franciscus Gasthuis (Other); Haaglanden Medical Centre (Other); Jeroen Bosch Ziekenhuis (Other); Maastricht University Medical Center (Other); Maxima Medical Center (Other); St. Antonius Hospital (Other); Laurentius ziekenhuis (Unknown); VieCuri Medical Centre (Other); NKI-AvL (Unknown); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Aarhus University Hospital (Other); Sheba Medical Center (Other Government); University of Florence (Other)
Responsible Party: Sponsor
Other Study IDs: W 21 04 00088
Record Dates: First submitted 2023-07-15; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mastectomy — Mastectomy as a surgical procedure for breast cancer (regardless of perioperative treatment).

SUMMARY:
Rationale:To improve the definition of the target volume for radiotherapy of the chestwall after different types of mastectomy, the exact localization of regions at risk for a local recurrence should be known. However, there are currently insufficient data in literature showing where local recurrences occur after different types of mastectomy.

Objective: The primary objective of the proposed study is to determine whether the spatial, location of a breast cancer recurrence after mastectomy, differs for different types of mastectomy.

Study design: Retrospective study evaluating spatial location and site of recurrences after mastectomy.

Study population: The investigators aim to include all breast cancer patients treated with mastectomy in the Netherlands between 2003- 2008, and known to have experienced a local recurrence as the first site of failure.

Primary endpoint: Spatial location of local recurrence (e.g., primary tumour bed, scar, skin, subcutaneous, nipple, areola, pectoral muscles).

DETAILED DESCRIPTION:
Rationale:To improve the definition of the target volume for radiotherapy of the chestwall after different types of mastectomy, the exact localization of regions at risk for a local recurrence should be known. However, there are currently insufficient data in literature showing where local recurrences occur after different types of mastectomy.

Objective: The primary objective of the proposed study is to determine whether the spatial, location of a breast cancer recurrence after mastectomy, differs for different types of mastectomy. Secondary objectives are to assess whether tumour characteristics (e.g., molecular subtypes, lymphangio/lymphovascular invasion) and treatment-related factors (e.g., PMRTwith or without bolus, radiation volumes, doses) influence the site of recurrence and spatial location.

Study design: Retrospective study evaluating spatial location and site of recurrences after mastectomy.

Study population: The investigators aim to include all breast cancer patients treated with mastectomy in the Netherlands between 2003- 2008, and known to have experienced a local recurrence as the first site of failure.

Primary endpoint: Primary endpoint: Spatial location of local recurrence (e.g., primary tumour bed, scar, skin, subcutaneous, nipple, areola, pectoral muscles).

Other study parameters: First descriptive statistics will be performed to investigate whether there is a relation between the localization of the recurrence and the type of mastectomy: modified radical mastectomy (MRM), skin-sparing mastectomy (SSM), nipple sparing mastectomy (NSM).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and more at the time of breast cancer diagnosis.
* Proven histology of first invasive breast cancer
* Mastectomy as a surgical procedure for breast cancer (regardless of perioperative treatment).
* Having a local recurrence, as primary event
* reast cancer diagnosis in the period 2003-2008.

Exclusion Criteria:

* Non-epithelial histology.
* Primary metastatic breast cancer.
* Mastectomy for breast cancer recurrence after earlier breast conserving therapy.
* Synchronous breast cancer.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: We aim to include all breast cancer patients treated with mastectomy in the Netherlands between 2003- 2008, and known to have experienced a local or regional recurrence or distant metastases as the first site of failure.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Spatial localisation of local recurrences | Up to 15 years after mastectomy
  The primary objective of the proposed study is to determine whether the spatial, location of a breast cancer recurrence after mastectomy, differs for different types of mastectomy.

SECONDARY OUTCOMES:
Influence of tumour characteristics on the site of recurrence and spatial location. | Up to 15 years after mastectomy
  Anaysis to assess whether tumour characteristics (e.g., molecular subtypes, lymphangio/lymphovascular invasion) influence the site of recurrence and spatial location.
Influence of treatment-related factors on the site of recurrence and spatial location. | Up to 15 years after mastectomy
  Anaysis to assess whether treatment-related factors (e.g., PMRT with or without bolus, radiation volumes, doses) influence the site of recurrence and spatial location.

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Boersma, Prof., Principal Investigator — Maastro
Locations (1):
- Maastro, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No